CLINICAL TRIAL: NCT01425476
Title: Breast Cancer Prevention Using Synergistic Prostaglandin Inhibitors (The Vitamin D/Celecoxib Study)
Brief Title: Changes in Breast Cancer Biomarkers Using Synergistic Prostaglandin Inhibitors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of North Dakota (Other)
Responsible Party: Principal Investigator, Edward Sauter, MD, PhD, M.H.A, The University of Texas Health Science Center at Tyler
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 200806
Record Dates: First submitted 2011-04-26; First posted 2011-08-30 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: breast; high risk women; biomarkers; vitamin D
MeSH Terms: conditions — Breast Neoplasms | interventions — Celecoxib; Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo & cholecalciferol 400 IU (Placebo Comparator): In this arm, the placebo is in place of celecoxib and the current RDA for cholecalciferol is used the control of the cholecalciferol higher dose.
  Interventions: Drug: Placebo; Drug: Cholecalciferol
- Placebo & cholecalciferol 2,000 IU (Active Comparator)
  Interventions: Drug: Placebo; Drug: Cholecalciferol
- celecoxib 400 mg & cholecalciferol 2,000 IU (Experimental)
  Interventions: Drug: Celecoxib; Drug: Cholecalciferol

INTERVENTIONS:
Drug: Celecoxib — Take one tablet from each bottle (one bottle containing either placebo/celecoxib and one bottle containing either cholecalciferol 400 IU or 2,000 IU) daily for 30 days.
  Other Names: celecoxib (Celebrex)
  Arms: celecoxib 400 mg & cholecalciferol 2,000 IU
Drug: Placebo — Take one tablet from each bottle (one bottle containing either placebo/celecoxib and one bottle containing either cholecalciferol 400 IU or 2,000 IU) daily for 30 days.
  Other Names: placebo (empty capsule inside an empty capsule)
  Arms: Placebo & cholecalciferol 2,000 IU; Placebo & cholecalciferol 400 IU
Drug: Cholecalciferol — Take one tablet from each bottle (one bottle containing either placebo/celecoxib and one bottle containing either cholecalciferol 400 IU or 2,000 IU) daily for 30 days.
  Other Names: cholecalciferol (Vitamin D)

SUMMARY:
This is a biomarker study with the goal of measuring changes in proteins and gene methylation. This study is not intended for use in diagnosing, mitigating, treating, curing, or preventing disease.

The purpose of this study is to determine if Vitamin D (cholecalciferol) alone and in combination with celecoxib (Celebrex, a non-steroidal anti-inflammatory drug, or NSAID), to decrease breast cancer risk by their effect on certain biological indicators (biomarkers) of breast cancer risk (called PGE2, COX-2, and 15-PGDH) and cell changes in the breast.

DETAILED DESCRIPTION:
This is a biomarker study with the goal of measuring changes in protein and RNA expression. This study is not intended for use in diagnosing, mitigating, treating, curing, or preventing disease.

66 women at high risk for breast cancer (gail risk >/= 1.66% for 5 year risk, or personal or family history)will be recruited and enrolled. 22 women will be randomized into each arm, with anticipation of 2 women in each group will not be evaluable, leaving 20 in each group for evaluation.

A combination of vitamin D and celecoxib act synergistically to decrease breast cancer risk by decreasing cell proliferation in the mammary epithelium through their action on prostaglandin synthesis and metabolism.

Specific Aims:

In women at increased breast cancer risk, determine the effect of vitamin D, with or without celecoxib, on

1. PG synthesis and metabolism, through the measurement of 15-PGDH, COX-2, and PGE2 in the breast

   Rationale: 1,25(OH)2D, the active form of vitamin D, has been shown in vitro to decrease PGE2 both by interfering with its production and by increasing its breakdown, leading to lower cell proliferation. Celecoxib potentiated the antiproliferative effect, allowing a much lower dose of each agent when used in combination than in isolation.
2. Proliferative activity in the breast, as measured by Mammary Ductoscopy (MD) cell morphology

   Rationale: Both MD and Nipple Aspirate Fluid (NAF) contain ductal epithelial cells, but MD samples contain more cells for cytologic review than NAF. Findings on MD cytology correlate with likelihood of breast cancer (2), NAF cytology relates to breast cancer risk and improves risk stratification (3), and bioactive food components can alter NAF cytology (4).
3. Circulating levels of 25(OH)D, 1,25(OH)2D, and celecoxib, and determine if the levels of these compounds correlate with response to markers of PG synthesis and metabolism or cell proliferation.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older
* Increased risk for breast cancer (demonstrated by strong family history [one 1st degree or two 2nd degree relatives], history of DCIS, IBC, or precancerous changes in breasts). OR Gail Model risk of developing IBC in a 5-year period of >1.66%
* Women with a history of breast cancer, must be free of disease and finished with treatment
* ECOG Performance Status score 0-1
* Premenopausal women must not be pregnant.

Exclusion Criteria:

* History of bilateral mastectomy, or bilateral breast irradiation
* Significant medical or psychiatric problems making the participant a poor candidate
* Evidence of excess use of narcotics or drug dependency
* Have been pregnant and lactating in the past 2 years
* Significant history of peptic ulcer disease or upper gastrointestinal bleeding
* History of severe congestive heart failure that requires hospitalization or intervention
* History of asthma requiring medication for treatment
* Allergy to sulfonamides or NSAID medications
* History of myocardial infarction or stroke
* Currently on Coumadin
* Currently on Tamoxifen (nolvadex),Evista (raloxifene), Femara (letrozole), Arimidex (anastrozole), or Aromasin (exemestane)
* Undergone prior subaeolar breast surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
PG synthesis and metabolism | approximately 30 days
  This will be measured from both baseline and completion samples.
  1. PG synthesis and metabolism, through the measurement of 15-PGDH, COX-2, and PGE2 in the breast
  Rationale: 1,25(OH)2D, the active form of vitamin D, has been shown in vitro to decrease PGE2 both by interfering with its production and by increasing its breakdown, leading to lower cell proliferation. Celecoxib potentiated the antiproliferative effect, allowing a much lower dose of each agent when used in combination than in isolation.

SECONDARY OUTCOMES:
Proliferative activity in the breast, as measured by MD cell morphology | approximately 30 days
  This will be measured from both baseline and completion samples.
  2. Proliferative activity in the breast, as measured by MD cell morphology
  Rationale: Both MD and NAF contain ductal epithelial cells, but MD samples contain more cells for cytologic review than NAF. Findings on MD cytology correlate with likelihood of breast cancer, NAF cytology relates to breast cancer risk and improves risk stratification, and bioactive food components can alter NAF cytology.
Circulating levels of 25(OH)D, 1,25(OH)2D, and celecoxib | approximately 30 days
  This will be measured from both baseline and completion samples.
  3. Circulating levels of 25(OH)D, 1,25(OH)2D, and celecoxib, and determine if the levels of these compounds correlate with response to markers of PG synthesis and metabolism or cell proliferation.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Sauter, MD, PhD, Principal Investigator — University of North Dakota
Locations (1):
- University of North Dakota, Grand Forks, North Dakota, United States